CLINICAL TRIAL: NCT05441254
Title: Camrelizumab Combined With Intraperitoneal Infusion of Nab-paclitaxel, Intravenous Chemotherapy and S-1 in the Treatment of Advanced Gastric Cancer With Peritoneal Metastasis：Single-arm, Prospective Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0627
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Stage IV Gastric Cancer With Metastasis
Keywords: Camrelizumab; Nab-paclitaxel; Peritoneal Metastasis; Intraperitoneal Infusion
MeSH Terms: interventions — camrelizumab; 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Camrelizumab: 200 mg, intravenous infusion, d1, q3w;
  Nab-paclitaxel: 130 mg/m2 intraperitoneal and 130 mg/m2 intravenously, d1, q3w;
  S-1: calculated based on body surface area Dosage, twice a day, orally, d1-d14, q3w;
  Interventions: Drug: Camrelizumab; Nab-paclitaxel; S-1

INTERVENTIONS:
Drug: Camrelizumab; Nab-paclitaxel; S-1 — Camrelizumab: 200 mg, intravenous infusion, d1, q3w;
  Nab-paclitaxel: 130 mg/m2 intraperitoneal and 130 mg/m2 intravenously, d1, q3w;
  S-1: calculated based on body surface area Dosage, twice a day, orally, d1-d14, q3w;
  The dosage can be adjusted according to the protocol according to the adverse reactions of subjects. Subjects will continue to take medication until completion of the prescribed course of treatment, disease progression, toxicity intolerance, withdrawal of Informed Consent Form, or termination in the investigator's judgment.
  Other Names: Arm PD-1

SUMMARY:
The purpose of this study was to evaluate the efficacy of camrelizumab combined with nab-paclitaxel intraperitoneal infusion, intravenous chemotherapy and S-1 in the treatment of advanced gastric cancer with peritoneal metastasis, so as to preliminarily explore the feasibility of the three-drug combination regimen in patients with gastric cancer with peritoneal metastasis and safety, and strive to maximize the benefits of different groups of people.

DETAILED DESCRIPTION:
The incidence of gastric cancer in China is high. Although the guidelines have recommended standard first and second-line chemotherapy, the survival rate of patients with advanced gastric cancer with peritoneal metastasis is still low.Nab-paclitaxel is a taxane drug, because of its binding to albumin, it does not need pretreatment before infusion, which is convenient for infusion, and has great application prospects in the treatment of advanced gastric cancer. There are positive expectations regarding the safety and efficacy of the combination. With the deepening of the understanding of the body's immune system and the rapid development of biotechnology, immunotherapy has become an important means of tumor treatment, and occupies an increasingly important position in the comprehensive tumor treatment system. At the same time, a number of studies have confirmed that camrelizumab combined with chemotherapy has a better therapeutic effect in gastric cancer, and the safety is tolerable.

In summary, how to improve the short-term and long-term efficacy of gastric cancer with peritoneal metastasis, while improving patient tolerance as much as possible and reducing adverse reactions, is an urgent problem to be solved. The purpose of this study was to evaluate the efficacy of camrelizumab combined with nab-paclitaxel intraperitoneal infusion, intravenous chemotherapy and S-1 in the treatment of advanced gastric cancer with peritoneal metastasis, so as to preliminarily explore the feasibility of the three-drug combination regimen in patients with gastric cancer with peritoneal metastasis and safety, and strive to maximize the benefits of different groups of people.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 years old ≤ age ≤ 75 years old, both male and female;
* 2.Pathology (including histology or cytology) confirmed gastric adenocarcinoma (papillary adenocarcinoma pap, tubular adenocarcinoma tub, mucinous adenocarcinoma muc, signet ring cell carcinoma sig, poorly differentiated adenocarcinoma por), and HER2- (HER2 Negative: IHC 0/1+ or IHC2+ but ISH negative);
* 3. Confirm the diagnosis of gastric cancer peritoneal metastasis by laparoscopy, laparotomy or imaging examination;
* 4. According to the RECIST1.1 standard, the patient has at least one target lesion with measurable diameter (the long diameter of the CT scan of the tumor lesion is ≥10mm, the short diameter of the CT scan of the lymph node lesion is ≥15mm, and the scan slice thickness is 5mm;)
* 5. The damage caused by the patient's other treatments has recovered, and the interval between receiving nitroso or mitomycin is ≥ 6 weeks; receiving other cytotoxic drugs, radiotherapy or surgery ≥ 4 weeks, and the wound has been completely healed;
* 6. ECOG PS: 0-2;
* 7.Expected survival ≥ 12 weeks;
* 8. The main organs function normally and meet the following criteria:

  1. Routine blood: (no blood transfusion within 14 days):

     1. HB≥100g/L,
     2. WBC≥3×109/L,
     3. ANC≥1.5×109/L,
     4. PLT≥100×109/L;
  2. Blood biochemistry:

     1. BIL <1.5ULN,
     2. ALT and AST <2.5ULN, GPT≤1.5×ULN,
     3. Serum Cr≤1ULN, endogenous creatinine clearance rate >60ml/min (Cockcroft-Gault formula),
     4. ALB≥30g/L;
* 9. Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the trial drug; for men, surgical sterilization or Agree to use an appropriate method of contraception during the trial and 8 weeks after the last administration of the trial drug;
* 10. Not participating in other clinical studies before and during treatment;
* 11. The patients voluntarily joined the study, signed the informed consent to participate in the experimental treatment, and agreed to participate in the observational study, with good compliance and cooperation with follow-up;
* 12. Has a quantifiable CT-PCI score.

Exclusion Criteria:

* 1. Patients who have previously received treatment with albumin-paclitaxel, Sigio, and camrelizumab; or patients who have previously received other immunotherapy (including other clinical research drugs) within 5 half-lives from the first study drug;
* 2. Concomitant Difficulties in swallowing, complete or incomplete gastrointestinal obstruction, active bleeding in the gastrointestinal tract, perforation, etc., etc.;
* 3. Participating in other clinical studies within 1 month before enrollment and the toxicity has not recovered;
* 4. There are a large number of Patients with ascites requiring frequent drainage that interferes with normal treatment;
* 5. Suffering from any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism , including but not limited to these diseases or syndromes); patients requiring no intervention in adulthood, except for vitiligo or cured childhood asthma/allergies; autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormones ; Type I diabetes mellitus using stable doses of insulin;
* 6. A history of immunodeficiency, including HIV test positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
* 7. Accompanied by severe heart, lung, liver and kidney diseases; neurological and mental diseases; jaundice or gastrointestinal obstruction and concomitant severe infection;
* 8. pregnant or breastfeeding women;
* 9. The presence of uncontrolled or symptomatic active central nervous system (CNS) metastases, which can manifest as clinical symptoms, cerebral edema, spinal cord compression meningitis, leptomeningeal disease, and/or progressive growth. CNS metastases are adequately treated, and neurological symptoms can return to baseline levels at least 2 weeks before enrollment (residual signs or symptoms associated with CNS treatment can be enrolled in the study). In addition, patients must discontinue corticosteroids or receive ≤10 mg/d of stable or tapered doses of prednisone (or equivalent doses of other corticosteroids) at least 2 weeks prior to enrollment;
* 10. Patients with grade I or above coronary heart disease, arrhythmia (including QTc interval prolongation > 450 ms in men, > 470 ms in women) and cardiac insufficiency;
* 11. Patients with clear gastrointestinal bleeding tendency, including the following conditions: Patients with locally active ulcer lesions, fecal occult blood (++), and a history of melena and hematemesis within 2 months; patients with abnormal coagulation function (INR>1.5, APTT>1.5 ULN);
* 12. The patient has uncontrolled cardiovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) ) Clinically significant supraventricular or ventricular arrhythmia without clinical intervention or still poorly controlled after clinical intervention;
* 13. History of interstitial lung disease (except radiation pneumonitis without hormone therapy), non-infectious pneumonia medical history;
* 14. Patients with positive urine protein (urinary protein test 2+ or above, or 24-hour urine protein quantification >1.0g);
* 15. Those who are allergic to the experimental drug or its excipients;
* 16. those who are considered unsuitable for inclusion by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 24 months
  Defined as the time from the date of informed consent to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  Defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Peritoneal Cancer Index (PCI) assessed on preoperative CT (CT-PCI) | 24 months

OTHER OUTCOMES:
Adverse event (AE) rate, serious adverse event (SAE) rate, etc | 24 months
  According to NCI CTC Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiao, Phd, Principal Investigator — Zhongshan Hospital Affiliated to Xiamen University